CLINICAL TRIAL: NCT05901493
Title: Improving the Retention of Speech-Perceptual Learning in Adults With and Without Language Disorder
Brief Title: Category Learning Retention in Adults With and Without Developmental Language Disorder
Acronym: Time2Learn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: Northeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1938428
Record Dates: First submitted 2023-05-19; First posted 2023-06-13 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Developmental Language Disorder; Adults Without Language Disorder
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of six training schedules to complete over 48 hours. All participants will complete the same amount of training. The investigators will examine retention of trained information at the end of the week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Blocked Evening Only Training (Experimental): One hour training in the evening, followed by a one hour training 24 hours later
  Interventions: Behavioral: Perceptual category training
- Distributed Evening Training (Experimental): One hour training in the evening, followed by a two 30 min trainings 12 and 24 hours later
  Interventions: Behavioral: Perceptual category training
- Blocked Evening-Morning Training (Experimental): One hour training in the evening, followed by a one hour training 12 hours later
  Interventions: Behavioral: Perceptual category training
- Blocked Morning Only Training (Experimental): One hour training in the morning, followed by a one hour training 24 hours later
  Interventions: Behavioral: Perceptual category training
- Distributed Morning Training (Experimental): One hour training in the morning, followed by a two 30 min trainings 12 and 24 hours later
  Interventions: Behavioral: Perceptual category training
- Blocked Morning-Evening Training (Experimental): One hour training in the morning, followed by a one hour training 12 hours later
  Interventions: Behavioral: Perceptual category training

INTERVENTIONS:
Behavioral: Perceptual category training — Participants complete a forced-choice categorization task with feedback, in order to learn difficult auditory and visual categories

SUMMARY:
Approximately 7% of the population experiences developmental language disorder (DLD), a language disorder with unclear causes. DLD affects communication beyond adolescence and poses challenges for education and career advancement due to difficulties in learning and memory. Recent research suggests that adults with DLD struggle with overnight memory consolidation, indicating a need for effective learning and memory support. This project aims to determine the optimal training schedule for perceptual memory retention in adults with and without DLD. The study involves recruiting 240 adults (120 with DLD, 120 without) for speech-perceptual training with different training schedules. The researchers predict that the manipulation of training schedules will interact with circadian preference and overnight consolidation, leading to the discovery of the best practice schedule for speech sound retention. Additionally, 300 more adults (150 with DLD, 150 without) will be recruited to investigate how optimal training schedules interact with reflexive and reflective learning strategies. The time course of learning and retention will be tracked during reflexive and reflective categorization training in six different training schedules.

DETAILED DESCRIPTION:
Developmental language disorder (DLD) describes the idiopathic disorder(s) of language that occurs in approximately 7% of the population. Although DLD is understudied in adulthood, it is clear that the communication challenges in DLD extend beyond adolescence. The barriers to educational and vocational achievement for adults with DLD include persistent difficulties in learning and memory. Recent work suggests that these difficulties with learning and memory include deficits in overnight memory consolidation. Thus, an effective support for learning and memory function in adults with DLD must include strategies for both overcoming initial challenges in learning, as well as in mitigating a deficit in consolidation of learned information. In this project, the investigators combine insights from the neurobiology of learning and memory, chronobiology, and speech perception, to determine the optimal training schedule for perceptual memory retention in adults with and without DLD. The investigators have two Aims in this project: First, the investigators will recruit 240 adults (120 with/120 without DLD) to participate in a speech-perceptual training to take place in one of six different training schedules over 24 hours. The investigators predict that our manipulation of training schedules will interact with circadian preference and timing relative to overnight consolidation, to allow the discovery of the optimal practice schedule for speech sound retention for adult learners with & without DLD. Under our second aim, the investigators will recruit an additional 300 adults (150 with/150 without DLD) in order to determine how optimal training schedules interact with reflexive and reflective learning strategies in adults with and without DLD. The investigators will achieve this aim by tracking the time course of learning and retention in adults participating in reflexive and reflective categorization training in one of six training schedules.

ELIGIBILITY:
Inclusion Criteria:

* native speakers of American English
* Grew up in a household in which only American English was spoken
* 18-55 years of age
* Typical vision & hearing
* (Aim 2) access to headphones/devices capable of accessing experiment script via internet
* Must meet criteria for Group membership as either TD or DLD

Exclusion Criteria:

* History of neurological disorders
* History of psychiatric disorders
* History of socio-emotional disorders
* On prescription medication(s) that alter sleep

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 540 (Estimated)
Dates: Start 2022-10-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Speech discrimination - behavior | 1 week
  Participants will be administered a short (approximately 4-minute) behavioral task. They will be exposed to two speech sounds, separated by a 1-second interval. Some sounds will begin with the dental stop consonant, and other sounds will begin with the retroflex stop consonant. Participants will be asked to decide if the two sounds they hear are the same or different. Accuracy will be converted to d-prime (a measure of signal detection). This d-prime score will be the primary behavioral outcome for speech discrimination.
category identification - behavior | 48 hours
  Participants will be administered a short (approximately 2 minutes) for each modality (auditory and visual). Participants will either hear (auditory - pure tone) or see (visual - gabor patch) a stimulus, and will need to choose which category the stimulus belongs to out of a choice of two. The percentage of trials that are answered correctly will be the primary behavioral outcome for auditory and visual category identification.

SECONDARY OUTCOMES:
Speech discrimination - Event-related potential of the electroencephalogram (ERP/EEG) | 1 event-related potential (ERP) session 1 week following training
  The investigators will fit the participant's head with a pre-positioned electrode cap, with electrolytic gel applied between the electrodes and the scalp. The participants will watch a silent movie while dental and retroflex speech tokens are presented in an oddball paradigm. The investigators will record the participants' electroencephalogram (EEG) while the auditory stimuli are presented. The EEG data will be segmented to examine the fluctuations in voltage recorded at the scalp (in milivolts) for a duration of one second after the onset of each stimulus. The segmented data will be averaged across dental trials, and across the retroflex trials. The resultant waveforms will be subtracted from one another. The peak of the deflection in the difference waveform found approximately 250miliseconds following stimulus onset is the mismatch negativity (MMN) component. The magnitude of the MMN component will be our primary outcome measure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Delaware, Newark, Delaware
  - Northeastern University, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
de-identified data will be uploaded to the Open Science Framework alongside publications to stem from data from this project
Supporting Information: Analytic Code
Time Frame: This data will be made available upon publication of the data, indefinitely